CLINICAL TRIAL: NCT06635629
Title: Phase II Prospective Evaluation of Desmopressin Stimulation Test Performance in ACTH-dependent Cushing s Syndrome
Brief Title: Desmopressin Stimulation Test Performance in ACTH-Dependent Cushing Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10001822; 001822-DK
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10-21

CONDITIONS: Cushing Syndrome
Keywords: desmopressin, Cushing syndrome, diagnosis
MeSH Terms: conditions — Cushing Syndrome; Disease | interventions — Deamino Arginine Vasopressin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Desmopressin 10 mcg Ad-lib fluid (Other): Desmopressin 10 mcg Ad-lib fluidHealthy volunteers only
  Interventions: Drug: Desmopressin
- Desmopressin 10 mcg NPO (Active Comparator): Desmopressin 10 mcg
  Interventions: Drug: Desmopressin
- Desmopressin NPO 4 mcg (Active Comparator): Desmopressin 4 mcg
  Interventions: Drug: Desmopressin
- Dexmopressin 10 mcg NPO + Dexamethasone (Active Comparator): Desmopressin 10 mcgDexamethasone 1 mg pretreatment
  Interventions: Drug: Desmopressin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Desmopressin — Stimulates ACTH release in Cushing disease
Drug: Dexamethasone — Inhibits ACTH release in Cushing disease and healthy volunteers
  Arms: Dexmopressin 10 mcg NPO + Dexamethasone

SUMMARY:
Background:

Cushing syndrome (CS) is a set of diseases that develop when the body produces too much adrenocorticotropic hormone (ACTH). ACTH stimulates the production of a hormone called cortisol. Excess cortisol can cause serious issues, such as diabetes, high blood pressure, weight gain, and mood changes. Diagnosing CS early can be difficult. One test used to diagnose CS, the desmopressin (Desmo) stimulation test (DesmoST), has not been studied in enough people to know how accurate it is.

Objective:

To find ways to improve the DesmoST. Researchers especially want to learn more about how well the DesmoST identifies people with specific ACTH CSs: Cushing disease (CD) and ectopic ACTH syndrome (EAS).

Eligibility:

People aged 18 to 70 years who have or may have CS, especially CD or EAS. Healthy volunteers are also needed.

Design:

Participants with CS will have 3 DesmoSTs at least 48 hours apart. The procedure for each is as follows:

They will limit their fluid intake the day before each test. They will have nothing to eat or drink for 12 hours before the test.

For 1 of the tests, they will take a pill that contains a hormone (dexamethasone). They will take it around 11 pm the day before the test.

Desmo is given through a tube attached to a needle inserted into a vein.

Blood will be drawn a total of 6 times before and after the desmo is given.

Healthy volunteers will have 4 DesmoSTs. These will be 2 to 14 days apart.

All participants will have follow-up visits 3 to 5 days after each test. These visits may be by phone.

DETAILED DESCRIPTION:
Study Description:

The goal of this study is to improve the diagnostic accuracy of the Desmopressin stimulation test (DesmoST) for three indications: to identify the etiology of ACTH-dependent Cushing syndrome (CS) as either Cushing Disease (CD) or Ectopic ACTH Syndrome (EAS), to discriminate between non-CS subjects (healthy controls and patients with pseudo-CS) and CD, and to identify CD in patients with cyclic hypercortisolism or recurrence. Test conditions include ad libitum water intake vs fluid restriction; increased glucocorticoid negative feedback (1 mg dexamethasone); and variable doses of desmopressin (4 mcg vs 10 mcg). We hypothesize that fluid restriction (via increased endogenous vasopressin levels), increased glucocorticoid negative feedback, and a lower dose of desmopressin improve specificity.

Objectives:

-Primary Objective:

To evaluate the hormonal response to desmopressin in subjects with ACTHdependent Cushing syndrome (CD and EAS) and non-CS subjects (healthy controls, pseudo-CS) under different conditions.

-Secondary Objective:

To evaluate the DesmoST performance (sensitivity, specificity, diagnostic accuracy) in identifying CD and distinguishing it from EAS and non-CS under different conditions.

-Exploratory Objectives:

To evaluate the ability of the DesmoST to identify CD in patients with cyclic hypercortisolism or postoperative recurrence; to evaluate whether Factor VIII is a biomarker for desmopressin action; and to explore the relationship between fluid status and response to desmopressin

Endpoints:

-Primary Endpoints:

Percentage change of peak ACTH and cortisol from baseline levels during the DesmoST under different conditions.

-Secondary Endpoints:

Cut-off points of relative ACTH and cortisol increase during the DesmoST that produce optimal diagnostic accuracy, once diagnostic information from other tests/imaging has been used to categorize subjects with suspected CS as having CD, EAS, or pseudo-CS.

-Exploratory Endpoints:

Percent change of peak ACTH and cortisol from baseline during the DesmoST in patients categorized as having cyclic hypercortisolism, postoperative recurrence, and fluid replete or restricted; the change in factor VIII levels after desmopressin administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged 18-70 years
* Agreement to adhere to Lifestyle Considerations throughout the study.
* Evidence of acceptable laboratory testing results within four weeks of the first test day, as shown by medical record review:

  * Hematocrit at entry >=33 %
  * Plasma sodium 136-145 mmol/L (unless taking a drug that can cause hyponatremia, see below) eGFR >=60 ml/min/1.73 sq.m, calculated based on serum creatinine
* For subjects taking any drug that could worsen hyponatremia, a normal plasma sodium (136-145 mmol/L) must have been obtained within seven days of the first test day.

In addition, an individual must meet all the criteria listed for their diagnostic group below, based on medical record review:

A. Patients with possible ACTH-dependent Cushing Syndrome (where the results of further work up will classify the patient as having CD, EAS or pseudo-CS):

1. A. Hypercortisolemia as evidenced by physician note or laboratory report: at least one screening modality (1 mg dexamethasone suppression test, 24-hour urinary free cortisol (UFC), bedtime or late night (2200h - 2359h) salivary or serum cortisol) within 4 weeks of screening. In patients suspected to have cyclic CS any previous abnormal result will suffice.
2. A. Normal or increased plasma ACTH (>20 pg/mL) as evidenced by physician note or laboratory report.

B. Patients with recurrent ACTH-dependent Cushing Syndrome (previous CD or EAS):

1B. Evidence of previous remission of CD or EAS after resection of a causative pituitary or ectopic tumor, evidence of current ACTH-dependent hypercortisolism, and willingness to undergo repeat surgery.

C. Healthy volunteers:

C1. In good general health as evidenced by medical history and physical examination; and in a stable state of health without ongoing acute/temporary illness per the clinical judgement of the investigator.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study, based on medical record review (possible Cushing syndrome patients) or a screening visit (healthy volunteers).

1. Inability to comply with all study procedures and visits
2. Inability of subject to understand or to sign a written informed consent document.
3. Known allergy/hypersensitivity to desmopressin.
4. Pregnancy or lactation, due to alterations in measured serum cortisol and lack of data on desmopressin safety.
5. A history of angina, significant coronary artery disease, congestive heart failure, or syndrome of inappropriate antidiuretic hormone secretion (SIADH), due to risk of fluid overload and/or hyponatremia.
6. Uncontrolled hypertension (blood pressure >150/95 mmHg) at screening and before desmopressin administration, due to risk of further increase if fluid overload occurs
7. Any condition that in the opinion of the Investigator would jeopardize the participant s appropriate participation in this study.
8. Current daily use of any of the following medications:

   * Drug used for the stimulation tests: Desmopressin.
   * Drugs that can suppress ACTH and cortisol test responses: Systemic glucocorticoids, including inhaled or topical formulations.
   * Vasopressors: phenylephrine, dopamine and vasopressin.
   * Drugs that interfere with desmopressin duration of action or potency: carbamazepine, lamotrigine, tolvaptan
9. Daily use of strong inducers of CYP3A4 (e.g. barbiturates, phenytoin, rifampin, rifabutin, rifapentine, carbamazapine, eslicarbazepine, primidone, cenobamate, Modafinil). Use of St John's wort or nafcillin within 14 days.
10. Initiation or dose increase within the past 14 days of drugs that can worsen hyponatremia: non-steroidal anti-inflammatory drugs (NSAIDs), loop diuretics (bumetanide, ethacrynic acid, furosemide, torsemide), chlorpromazine, chlorpropamide, cisplatin, monoamine oxidase inhibitors (MAOI), opiate agonists, oxybutynin, selective serotonin reuptake inhibitors (SSRI), vincristine, tricyclic antidepressants (TCAs)
11. Chronic enhanced hydration (estimated as >4 liters) to supplement mealtime fluid intake.
12. Any contraindication to intravenous catheter use.
13. Previous participation in this protocol.
14. History of hemophilia of any type.
15. Any hematology or chemistry screening laboratory value drawn at screening that the Investigator determines is clinically significant for exclusion.

Condition-specific exclusions will also apply to each subject group as follows:

A.Patients with possible ACTH-dependent Cushing Syndrome:

1. A. Use of medications that block glucocorticoid production (ketoconazole, levoketoconazole, metyrapone, osilodrostat) within the past two weeks, if normal cortisol is achieved. If hypercortisolism persists despite the use of these medications, as evidenced by an elevated 24-hour urinary free cortisol (UFC) or late night (2200h - 2359h) salivary or serum cortisol within two weeks of the first desmopressin test, the medication(s) may be continued until 48 hours before the first desmopressin test.
2. A. Use of the adrenolytic mitotane at any point, due to its prolonged half-life.
3. A. Use of medications that block glucocorticoid action or ACTH release within the past two weeks - mifepristone, cabergoline, octreotide (subcutaneous), pasireotide (subcutaneous), megestrol acetate, other synthetic glucocorticoids (except for topical or inhaled agents and single doses of oral dexamethasone for diagnostic testing within the past 48 hours)
4. A. Use of intramuscular long-acting forms of octreotide or pasireotide within the past 4 months.
5. A. Treatment of diabetes insipidus.

B. Healthy volunteers:

1. B. Use of oral, injectable, or inhaled glucocorticoids (unless intermittent, for symptomatic asthma) within the last year. Use of topical non-hydrocortisone containing potent glucocorticoids on more than 36 square inches in the last six months.
2. B. Hemoglobin A1c >= 6.5% on screening labs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
ACTH and cortisol responses | -5, 0, 15, 30, 45 and 60 minutes
  Percent change from mean baseline values (-5, 0 minutes) at all combinations of dose dose timepoints

SECONDARY OUTCOMES:
Diagnostic accuracy, specificity, sensitivity of cortisol and ACTH measurements in response to desmopressin | -5, 0, 15, 30, 45 and 60 minutes
  ROC curve % +/- 95% Confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data appearing in publications will be shared.
Supporting Information: Analytic Code
Time Frame: Beginning 6 months after publication
Access Criteria: The PI will review requests for data sharing. Data will shared for scientific analysis

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001822-DK.html